CLINICAL TRIAL: NCT00090285
Title: An Investigational Vaccine in Reducing the Incidence of Anogenital Warts in Young Men
Brief Title: An Investigational Study of Gardasil™ (qHPV Vaccine) in Reducing the Incidence of Anogenital Warts in Young Men (V501-020)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-020; Formerly-0904HPVHMES; 2004_103; 2004-002945-10 (EudraCT Number); V501-020 (Other: Merck Protocol Number)
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Condylomata Acuminata
Keywords: anogenital warts
MeSH Terms: conditions — Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Vaccines, Synthetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- qHPV Vaccine (Experimental): The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time participants received qHPV vaccination at Day 1, Month 2 and Month 6. Follow-up for the Base Study encompassed Month 7 through Month 36.
  Interventions: Biological: (Gardasil™) human papillomavirus (types 6, 11, 16, 18) recombinant vaccine
- Placebo (Placebo Comparator): The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time participants received placebo at Day 1, Month 2 and Month 6. Follow-up for the Base Study encompassed Month 7 through Month 36.
  Interventions: Biological: Comparator: placebo (unspecified)

INTERVENTIONS:
Biological: (Gardasil™) human papillomavirus (types 6, 11, 16, 18) recombinant vaccine — 0.5 mL intramuscular injection in the deltoid muscle at Day 1, Month 2, and Month 6 in the Base Study
  Other Names: qHPV; V501
  Arms: qHPV Vaccine
Biological: Comparator: placebo (unspecified) — 0.5 mL intramuscular injection in the deltoid muscle at Day 1, Month 2, and Month 6 in the Base Study
  Arms: Placebo

SUMMARY:
This study was conducted to demonstrate that Gardasil™ (quadrivalent human papillomavirus [qHPV] vaccine) 1) is well tolerated in young men, 2) reduces incidence of external genital lesions in young men, 3) reduces the incidence of anal intraepithelial neoplasia (AIN) or anal cancer in men having sex with men (MSM), and 4) reduces incidence of Human Papillomavirus (HPV) infection in young men. In the 7-month Base Study participants received randomly assigned qHPV vaccine or placebo at Day 1, Month 2, and Month 6. Base Study follow-up continued through Month 36. In Extension 1 (EXT1), participants who received placebo or an incomplete qHPV vaccine regimen in the Base Study were offered qHPV vaccine. Participants were followed in EXT1 for 7 months. In Extension 2 [LTFU (EXT2)], long-term effectiveness, immunogenicity, and safety of qHPV vaccine were followed up to 10 years following study enrollment. Participants who received ≥1 dose of qHPV vaccine in the Base Study or EXT1 were eligible to enroll in LTFU (EXT2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy heterosexual males between the ages of 16 years and 23 years and 364 days. Healthy men having sex with men (MSM) between the ages of 16 years and 26 years and 364 days.
* No clinical evidence of genital lesions suggesting sexually-transmitted disease, and no history of anogenital warts
* Additional criteria will be discussed with you by the physician

Exclusion Criteria:

* Concurrently enrolled in a clinical study involving collection of genital specimens
* History of known prior vaccination with an HPV vaccine
* Received an inactivated vaccine within 14 days or a live virus vaccine within 21 days prior to enrollment
* History of a severe allergic reaction that required medical intervention
* Received any immune globulin or blood-derived products within 6 months prior to the first study injection
* History of splenectomy, immune disorders, or receiving immunosuppressives
* Immunocompromised or diagnosed with HIV infection
* Known thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections
* History of recent or ongoing alcohol or drug abuse

Ages: 16 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4065 (Actual)
Dates: Start 2004-09-03 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinicaltrials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Broshkevitch CJ, Giuliano AR, Palefsky JM, Nahhas G, Goldstone SE, Dubin B, Saah A, Luxembourg A, Velicer C, Tota JE. Assessment of Concordant Human Papillomavirus Infection With 9-Valent Vaccine Types Across Anogenital Sites in Young Men. J Infect Dis. 2025 Dec 16:jiaf564. doi: 10.1093/infdis/jiaf564. Online ahead of print. PMID 41400842
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Giuliano AR, Palefsky JM, Goldstone SE, Dubin B, Saah A, Luxembourg A, Velicer C, Tota JE. High Risk of New HPV Infection Acquisition Among Unvaccinated Young Men. J Infect Dis. 2024 Mar 14;229(3):707-718. doi: 10.1093/infdis/jiad485. PMID 38012959
- [Derived] Goldstone SE, Giuliano AR, Palefsky JM, Lazcano-Ponce E, Penny ME, Cabello RE, Moreira ED Jr, Baraldi E, Jessen H, Ferenczy A, Kurman R, Ronnett BM, Stoler MH, Bautista O, Das R, Group T, Luxembourg A, Zhou HJ, Saah A. Efficacy, immunogenicity, and safety of a quadrivalent HPV vaccine in men: results of an open-label, long-term extension of a randomised, placebo-controlled, phase 3 trial. Lancet Infect Dis. 2022 Mar;22(3):413-425. doi: 10.1016/S1473-3099(21)00327-3. Epub 2021 Nov 12. PMID 34780705
- [Derived] Tota JE, Giuliano AR, Goldstone SE, Dubin B, Saah A, Luxembourg A, Velicer C, Palefsky JM. Anogenital Human Papillomavirus (HPV) Infection, Seroprevalence, and Risk Factors for HPV Seropositivity Among Sexually Active Men Enrolled in a Global HPV Vaccine Trial. Clin Infect Dis. 2022 Apr 9;74(7):1247-1256. doi: 10.1093/cid/ciab603. PMID 34265048
- [Derived] Doshi P, Bourgeois F, Hong K, Jones M, Lee H, Shamseer L, Spence O, Jefferson T. Adjuvant-containing control arms in pivotal quadrivalent human papillomavirus vaccine trials: restoration of previously unpublished methodology. BMJ Evid Based Med. 2020 Dec;25(6):213-219. doi: 10.1136/bmjebm-2019-111331. Epub 2020 Mar 17. PMID 32184277
- [Derived] Goldstone SE, Jessen H, Palefsky JM, Giuliano AR, Moreira ED Jr, Vardas E, Aranda C, Hillman RJ, Ferris DG, Coutlee F, Marshall JB, Vuocolo S, Haupt RM, Guris D, Garner E. Quadrivalent HPV vaccine efficacy against disease related to vaccine and non-vaccine HPV types in males. Vaccine. 2013 Aug 20;31(37):3849-55. doi: 10.1016/j.vaccine.2013.06.057. Epub 2013 Jul 2. PMID 23831322
- [Derived] Palefsky JM, Giuliano AR, Goldstone S, Moreira ED Jr, Aranda C, Jessen H, Hillman R, Ferris D, Coutlee F, Stoler MH, Marshall JB, Radley D, Vuocolo S, Haupt RM, Guris D, Garner EI. HPV vaccine against anal HPV infection and anal intraepithelial neoplasia. N Engl J Med. 2011 Oct 27;365(17):1576-85. doi: 10.1056/NEJMoa1010971. PMID 22029979
- [Derived] Giuliano AR, Palefsky JM, Goldstone S, Moreira ED Jr, Penny ME, Aranda C, Vardas E, Moi H, Jessen H, Hillman R, Chang YH, Ferris D, Rouleau D, Bryan J, Marshall JB, Vuocolo S, Barr E, Radley D, Haupt RM, Guris D. Efficacy of quadrivalent HPV vaccine against HPV Infection and disease in males. N Engl J Med. 2011 Feb 3;364(5):401-11. doi: 10.1056/NEJMoa0909537. PMID 21288094

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4164 participants were screened and 4065 were randomized
Groups:
- qHPV Vaccine in Base Study: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time participants received quadrivalent human papillomavirus (qHPV) vaccination at Day 1, Month 2 and Month 6.
  Follow-up for the Base Study encompassed Month 7 through Month 36.
- Placebo in Base Study: The Vaccination Period for the Base study encompassed Day 1 through Month 7, during which time participants received placebo at Day 1, Month 2 and Month 6.
  Follow-up for the Base Study encompassed Month 7 through Month 36.
- EXT1: Placebo in Base Study: Participants in the placebo arm in the base study were offered 3 doses of open-label qHPV vaccine at Extension 1 (EXT1) Day 1, Month 2 and Month 6.
  Participants were followed to EXT1 Month 7.
- EXT1: Incomplete qHPV Regimen in Base Study: Participants who received only 1 dose of qHPV vaccine in the Base Study were offered a complete 3-dose qHPV vaccine regimen (administered at EXT1 Day 1, Month 2 and Month 6). Participants who received only 2 doses of qHPV vaccine in the Base Study were offered a single additional dose of qHPV vaccine (administered at EXT1 Day 1).
  Participants were followed to EXT1 Month 7.
- LTFU (EXT2): Early Vaccination Group: Participants received ≥1 dose of qHPV vaccine in Base Study and were followed up to a total of 10 years after their first dose of qHPV vaccine. No vaccinations were administered during Long-term Follow-up (LTFU) (EXT2).
- LTFU (EXT2): Catch-up Vaccination Group: Participants received placebo in Base Study and qHPV vaccine in EXT1 and were followed up to a total of 7 years after their first dose of qHPV vaccine. No vaccinations were administered during LTFU (EXT2).
Period: Base Study Vaccination Period
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | EXT1: Placebo in Base Study | EXT1: Incomplete qHPV Regimen in Base Study | LTFU (EXT2): Early Vaccination Group | LTFU (EXT2): Catch-up Vaccination Group
Started | 2032 | 2033 | 0 | 0 | 0 | 0
Vaccinated | 2025 | 2030 | 0 | 0 | 0 | 0
Completed | 1818 | 1814 | 0 | 0 | 0 | 0
Not Completed | 214 | 219 | 0 | 0 | 0 | 0
Not completed — Randomized Not Vaccinated | 7 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 111 | 112 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 64 | 69 | 0 | 0 | 0 | 0
Not completed — Uncooperative | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Moved | 20 | 21 | 0 | 0 | 0 | 0
Not completed — Site Terminated | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Subject Incarcerated | 2 | 2 | 0 | 0 | 0 | 0
Not completed — HIV positive | 1 | 1 | 0 | 0 | 0 | 0
Period: Base Study Follow-up Period
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | EXT1: Placebo in Base Study | EXT1: Incomplete qHPV Regimen in Base Study | LTFU (EXT2): Early Vaccination Group | LTFU (EXT2): Catch-up Vaccination Group
Started | 1822 (4 subjects who did not receive 3 doses of vaccine in base study continued into the Follow-up Period) | 1821 (7 subjects who did not receive 3 doses of placebo in base study continued into the Follow-up Period) | 0 | 0 | 0 | 0
Completed | 1487 | 1479 | 0 | 0 | 0 | 0
Not Completed | 335 | 342 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 10 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 232 | 226 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 53 | 64 | 0 | 0 | 0 | 0
Not completed — Moved | 41 | 36 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Uncooperative | 3 | 4 | 0 | 0 | 0 | 0
Not completed — Subject Incarcerated | 0 | 2 | 0 | 0 | 0 | 0
Period: Extension 1
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | EXT1: Placebo in Base Study | EXT1: Incomplete qHPV Regimen in Base Study | LTFU (EXT2): Early Vaccination Group | LTFU (EXT2): Catch-up Vaccination Group
Started | 0 | 0 | 1098 (Participation in EXT1 was voluntary; not all participants eligible for EXT1 enrolled.) | 16 (Participation in EXT1 was voluntary; not all participants eligible for EXT1 enrolled.) | 0 | 0
Completed | 0 | 0 | 1041 | 15 | 0 | 0
Not Completed | 0 | 0 | 57 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 35 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 13 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Moved | 0 | 0 | 3 | 0 | 0 | 0
Period: Long-term Follow-up (EXT2)
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | EXT1: Placebo in Base Study | EXT1: Incomplete qHPV Regimen in Base Study | LTFU (EXT2): Early Vaccination Group | LTFU (EXT2): Catch-up Vaccination Group
Started | 0 | 0 | 0 | 0 | 936 (Not all eligible participants enrolled in LTFU (EXT2)) | 867 (Not all eligible participants enrolled in LTFU (EXT2))
Completed | 0 | 0 | 0 | 0 | 709 | 664
Not Completed | 0 | 0 | 0 | 0 | 227 | 203
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 156 | 143
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 60 | 53
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- qHPV Vaccine in Base Study: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time participants received qHPV vaccination at Day 1, Month 2 and Month 6.
  Follow-up for the Base Study encompassed Month 7 through Month 36.
- Total: Total of all reporting groups
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study | Total
Number analyzed (Participants) | 2032 | 2033 | 4065
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.6 (2.0) | 20.5 (2.0) | 20.5 (2.0)
Age, Continuous [Median (Full Range); unit: Years] — Although the upper age limit for this study was 26 years old, one subject age 27 was randomized into the study.
  Years | 20 [16 to 26] | 20 [15 to 27] | 20 [15 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2032 | 2033 | 4065
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 201 | 205 | 406
  Black | 405 | 400 | 805
  Hispanic American | 412 | 423 | 835
  Native American | 1 | 2 | 3
  White | 719 | 712 | 1431
  Multi-Racial | 291 | 283 | 574
  Indian (subcontinent) | 1 | 8 | 9
  Polynesian | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Base Study: Incidence of Human Papillomavirus (HPV) Type 6/11/16/18-related External Genital Warts, Penile/Perianal/Perineal Intraepithelial Neoplasia (PIN), Penile, Perianal or Perineal Cancer
Description: Participants with HPV 6/11/16/18-related external genital warts, penile/perianal/perineal intraepithelial neoplasia (PIN), penile, perianal or perineal cancer per 100 person-years of follow-up was assessed.
Time Frame: Base study: through Month 36
Population: Participants must have received 3 doses of qHPV vaccine or placebo, have no protocol violations that could interfere with the effects of the vaccine, be seronegative at Day 1 and PCR negative Day 1 through Month 7 for the relevant HPV type, and must provide data after Month 7.
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1394 | 1404
Incidence per 100 person-years | 0.1 | 1.0
Statistical Analysis 1: Comparison: qHPV Vaccine in Base Study vs Placebo in Base Study; Test type: Superiority or Other; Risk Difference (RD) = 90.6, 95% CI [70.1 to 98.2] — Confidence Interval (CI) based on binomial tail probabilities and not from a dispersion parameter

2. Primary Outcome: Overall Study: Incidence of HPV Type 6/11-related Genital Warts
Description: Incidence of HPV Type 6/11-related genital warts is expressed as events per 10,000 person-years of follow-up.
Time Frame: Up to 10 years after the first dose of qHPV vaccine
Population: Participants must have received 3 doses of qHPV vaccine, have no protocol violations that could interfere with the effects of the vaccine, be seronegative at Day 1 and PCR negative Day 1 through Month 7 for the relevant HPV type, and must provide data after Month 7. This endpoint applied only to participants in the Base Study qHPV vaccine group.
Measure: Number (95% Confidence Interval); unit: Incidence per 10,000 person-years
Groups:
- qHPV Vaccine in Base Study: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time participants received qHPV vaccination at Day 1, Month 2 and Month 6.
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 1243
Incidence per 10,000 person-years | 4.3 [0.9 to 12.5]

3. Primary Outcome: Overall Study: Incidence of HPV Type 6/11/16/18-related External Genital Warts, PIN, Penile, Perianal or Perineal Cancer
Description: Incidence of HPV Type 6/11/16/18-related external genital warts, PIN, penile, perianal or perineal cancer is expressed as events per 10,000 person-years of follow-up.
Time Frame: Up to 10 years after the first dose of qHPV vaccine
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Incidence per 10,000 person-years
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 1395
Incidence per 10,000 person-years | 3.8 [0.8 to 11.1]

4. Primary Outcome: Overall Study: Incidence of HPV Type 6/11/16/18-related Anal Intraepithelial Neoplasia (AIN) and Anal Cancer
Description: Incidence of HPV Type 6/11/16/18-related AIN and anal cancer is expressed as events per 10,000 person-years of follow-up. MSM is men having sex with men.
Time Frame: Up to 10 years after the first dose of qHPV vaccine
Population: Participants must have received 3 doses of qHPV vaccine, have no protocol violations that could interfere with the effects of the vaccine, be seronegative at Day 1 and PCR negative Day 1 through Month 7 for the relevant HPV type, and must provide data after Month 7. This endpoint applied only to MSM in the Base Study qHPV vaccine group.
Measure: Number (95% Confidence Interval); unit: Incidence per 10,000 person-years
Groups:
- MSM qHPV Vaccine in Base Study: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time participants received qHPV vaccination at Day 1, Month 2 and Month 6.
  Follow-up for the Base Study encompassed Month 7 through Month 36.
Arm/Group | MSM qHPV Vaccine in Base Study
Number analyzed (Participants) | 194
Incidence per 10,000 person-years | 69.3 [25.4 to 150.8]

5. Primary Outcome: Base Study: Number of Participants With Severe Injection Site Adverse Experiences (AEs)
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the SPONSOR'S product, is also an adverse experience. A severe AE is incapacitating with inability to work or do usual activities.
Time Frame: Base study: through Day 5 after any vaccination
Population: The analysis population included all vaccinated participants excluding 6 participants who received non-compliant mixed regimens of qHPV vaccine and placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study
Number analyzed (Participants) | 2020 | 2029
Participants | 25 | 20

6. Primary Outcome: Base Study: Number of Participants With Vaccine-Related Serious Adverse Events (SAEs)
Description: A serious adverse event is an AE that 1) results in death, 2) is life threatening, 3) results in persistent or significant disability or incapacity, 4) results in or prolongs an existing hospitalization, 5) is a congenital anomaly or birth defect, 6) is a cancer, 7) is an overdose, or 8) based on appropriate medical judgment may jeopardize the participant and may require medical or surgical intervention. A vaccine-related AE is one deemed to be possibly, probably or definitely related to study vaccine by the investigator.
Time Frame: Base study: through Month 36
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- qHPV Vaccine: Base Study and Followup: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time participants received qHPV vaccination at Day 1, Month 2 and Month 6.
  Follow-up for the base study encompassed Month 7 through Month 36. The at-risk population was participants who received ≥ 1 qHPV vaccination in the base study.
- Placebo: Base Study and Followup: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time participants received placebo at Day 1, Month 2 and Month 6.
  Follow-up for the base study encompassed Month 7 through Month 36. The at-risk population was participants who received ≥ 1 placebo injection in the base study.
Arm/Group | qHPV Vaccine: Base Study and Followup | Placebo: Base Study and Followup
Number analyzed (Participants) | 2020 | 2029
Participants | 0 | 0

7. Primary Outcome: LTFU (EXT2): Number of Participants With Vaccine-Related SAEs
Description: An SAE is an AE that 1) results in death, 2) is life threatening, 3) results in persistent or significant disability or incapacity, 4) results in or prolongs an existing hospitalization, 5) is a congenital anomaly or birth defect, 6) is a cancer, 7) is an overdose, or 8) based on appropriate medical judgment may jeopardize the participant and may require medical or surgical intervention. A vaccine-related AE is one deemed to be possibly, probably or definitely related to study vaccine by the investigator.
Time Frame: LTFU (EXT2): Early Vaccination Group: up to 12 years after last dose of qHPV vaccine; LTFU (EXT2) Catch-up Vaccination Group: up to 7 years after last dose of qHPV vaccine
Population: The population analyzed was all randomized participants receiving at least 1 dose of qHPV vaccine in the Base Study or EXT1 and enrolled in LTFU (EXT2).
Measure: Count of Participants; unit: Participants
Arm/Group | LTFU (EXT2): Early Vaccination Group | LTFU (EXT2): Catch-up Vaccination Group
Number analyzed (Participants) | 936 | 867
Participants | 0 | 0

8. Primary Outcome: LTFU (EXT2): Number of Participants Who Died
Description: The number of participants who died was assessed.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | LTFU (EXT2): Early Vaccination Group | LTFU (EXT2): Catch-up Vaccination Group
Number analyzed (Participants) | 936 | 867
Participants | 5 | 2

9. Other Pre Specified Outcome: Base Study: Substudy to Evaluate the Incidence of HPV 6/11/16/18-related Anal Intraepithelial Neoplasia (AIN) and Anal Cancer in Men Having Sex With Men (MSM)
Description: Participants with HPV 6/11/16/18-related AIN or anal cancer per 100 person-years of follow-up was assessed.
Time Frame: Base study: through Month 36
Population: Only a subset of participants was included for this sub-study. Participants must have received 3 doses of qHPV vaccine or placebo, have no protocol violations that could interfere with the effects of the vaccine, be seronegative at Day 1 and PCR negative Day 1 through Month 7 for the relevant HPV type, and must provide data after Month 7.
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study
Number analyzed (Participants) | 194 | 208
Incidence per 100 person-years | 1.3 | 5.8
Statistical Analysis 1: Comparison: qHPV Vaccine in Base Study vs Placebo in Base Study; Test type: Superiority or Other; Risk Difference (RD) = 77.5, 95% CI [39.6 to 93.3]

10. Secondary Outcome: Base Study: Incidence of HPV 6/11/16/18-related Persistent Infection
Description: Participants with HPV Type 6/11/16/18-related persistent infection per 100 person-years of follow-up was assessed.
Time Frame: Base study: through Month 36
Population: as for outcome 1
Measure: Number; unit: Infection per 100 person-years
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1390 | 1402
Infection per 100 person-years | 0.7 | 4.8
Statistical Analysis 1: Comparison: qHPV Vaccine in Base Study vs Placebo in Base Study; Test type: Superiority or Other; Risk Difference (RD) = 85.5, 95% CI [77.0 to 91.3] — CI based on binomial tail probabilities and not from a dispersion parameter. Hochberg multiplicity adjustment applied to the CI

11. Secondary Outcome: Base Study: Incidence of HPV 6/11/16/18-related Deoxyribonucleic Acid (DNA) Detection
Description: Participants with HPV 6/11/16/18-related DNA detection per 100 person-years of follow-up was assessed.
Time Frame: Base study: through Month 36
Population: as for outcome 1
Measure: Number; unit: Detection per 100 person-years
Arm/Group | qHPV Vaccine in Base Study | Placebo in Base Study
Number analyzed (Participants) | 1390 | 1402
Detection per 100 person-years | 5.3 | 10.7
Statistical Analysis 1: Comparison: qHPV Vaccine in Base Study vs Placebo in Base Study; Test type: Superiority or Other; Risk Difference (RD) = 51.0, 95% CI [40.3 to 59.9] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Geometric Mean Titers to HPV Types 6, 11, 16, and 18 at Month 7 Assessed by Competitive Luminex Immunoassay (cLIA)
Description: Antibodies to HPV types were measured using cLIA. Antibody titers were expressed as cLIA milli Merck units/mL (cLIA mMU/mL).
Time Frame: Month 7
Population: All participants who 1) were seronegative at Day 1 and PCR negative Day 1 through Month 7 for the relevant HPV type, 2) received all 3 vaccinations, and 3) did not have protocol deviations that could interfere with the effects of the vaccine. Immunogenicity was assessed only for participants who received qHPV vaccine in the Base Study.
Measure: Geometric Mean (95% Confidence Interval); unit: cLIA mMU/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
cLIA mMU/mL
  HPV Type 6: number analyzed (Participants) | 1090
  HPV Type 6 | 447.7 [415.9 to 481.9]
  HPV Type 11: number analyzed (Participants) | 1090
  HPV Type 11 | 624.4 [588.4 to 662.6]
  HPV Type 16: number analyzed (Participants) | 1133
  HPV Type 16 | 2406.1 [2245.0 to 2578.8]
  HPV Type 18: number analyzed (Participants) | 1173
  HPV Type 18 | 402.8 [373.9 to 433.9]

13. Secondary Outcome: Geometric Mean Titers to HPV Types 6, 11, 16, and 18 at Month 36 Assessed by cLIA
Description: as for outcome 12
Time Frame: Month 36
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: cLIA mMU/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
cLIA mMU/mL
  HPV Type 6: number analyzed (Participants) | 845
  HPV Type 6 | 71.5 [66.7 to 76.7]
  HPV Type 11: number analyzed (Participants) | 845
  HPV Type 11 | 82.5 [77.0 to 88.5]
  HPV Type 16: number analyzed (Participants) | 875
  HPV Type 16 | 293.6 [271.6 to 317.4]
  HPV Type 18: number analyzed (Participants) | 904
  HPV Type 18 | 33.2 [30.2 to 36.4]

14. Secondary Outcome: Geometric Mean Titers to HPV Types 6, 11, 16, and 18 at Month 72 Assessed by cLIA
Description: as for outcome 12
Time Frame: Month 72
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: cLIA mMU/mL
Groups:
- qHPV Vaccine in Base Study: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time participants received qHPV vaccination at Day 1, Month 2 and Month 6.
  Follow-up for the Base Study was through Month 36 and for LTFU (EXT2) was through Month 120.
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
cLIA mMU/mL
  HPV Type 6: number analyzed (Participants) | 575
  HPV Type 6 | 57.2 [52.3 to 62.5]
  HPV Type 11: number analyzed (Participants) | 575
  HPV Type 11 | 62.1 [56.7 to 68.1]
  HPV Type 16: number analyzed (Participants) | 609
  HPV Type 16 | 249.4 [225.6 to 275.8]
  HPV Type 18: number analyzed (Participants) | 633
  HPV Type 18 | 25.9 [23.2 to 28.9]

15. Secondary Outcome: Geometric Mean Titers to HPV Types 6, 11, 16, and 18 at Month 120 Assessed by cLIA
Description: as for outcome 12
Time Frame: Month 120
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: cLIA mMU/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
cLIA mMU/mL
  HPV Type 6: number analyzed (Participants) | 374
  HPV Type 6 | 49.4 [44.1 to 55.4]
  HPV Type 11: number analyzed (Participants) | 374
  HPV Type 11 | 38.7 [34.5 to 43.5]
  HPV Type 16: number analyzed (Participants) | 393
  HPV Type 16 | 182.9 [161.4 to 207.3]
  HPV Type 18: number analyzed (Participants) | 408
  HPV Type 18 | 17.6 [15.5 to 19.9]

16. Secondary Outcome: Percentage of Participants Seropositive for HPV Type 6, 11, 16, and 18 at Month 7 Assessed by cLIA
Description: Antibodies to HPV types were measured using cLIA. Thresholds for seropositive were ≥20, 16, 20, and 24 cLIA mMU/mL for HPV Types 6, 11, 16, and 18, respectively.
Time Frame: Month 7
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
Percentage of participants
  HPV Type 6: number analyzed (Participants) | 1090
  HPV Type 6 | 98.9 [98.1 to 99.4]
  HPV Type 11: number analyzed (Participants) | 1090
  HPV Type 11 | 99.2 [98.4 to 99.6]
  HPV Type 16: number analyzed (Participants) | 1133
  HPV Type 16 | 98.8 [97.9 to 99.3]
  HPV Type 18: number analyzed (Participants) | 1173
  HPV Type 18 | 97.4 [96.3 to 98.2]

17. Secondary Outcome: Percentage of Participants Seropositive for HPV Type 6, 11, 16, and 18 at Month 36 Assessed by cLIA
Description: as for outcome 16
Time Frame: Month 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
Percentage of participants
  HPV Type 6: number analyzed (Participants) | 845
  HPV Type 6 | 88.9 [86.6 to 90.9]
  HPV Type 11: number analyzed (Participants) | 845
  HPV Type 11 | 94.0 [92.1 to 95.5]
  HPV Type 16: number analyzed (Participants) | 875
  HPV Type 16 | 97.9 [96.8 to 98.8]
  HPV Type 18: number analyzed (Participants) | 904
  HPV Type 18 | 57.1 [53.8 to 60.3]

18. Secondary Outcome: Percentage of Participants Seropositive for HPV Type 6, 11, 16, and 18 at Month 72 Assessed by cLIA
Description: as for outcome 16
Time Frame: Month 72
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
Percentage of participants
  HPV Type 6: number analyzed (Participants) | 575
  HPV Type 6 | 84.3 [81.1 to 87.2]
  HPV Type 11: number analyzed (Participants) | 575
  HPV Type 11 | 88.0 [85.1 to 90.5]
  HPV Type 16: number analyzed (Participants) | 609
  HPV Type 16 | 97.0 [95.4 to 98.2]
  HPV Type 18: number analyzed (Participants) | 633
  HPV Type 18 | 49.6 [45.6 to 53.6]

19. Secondary Outcome: Percentage of Participants Seropositive for HPV Type 6, 11, 16, and 18 at Month 120 Assessed by cLIA
Description: as for outcome 16
Time Frame: Month 120
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
Percentage of participants
  HPV Type 6: number analyzed (Participants) | 374
  HPV Type 6 | 79.1 [74.7 to 83.2]
  HPV Type 11: number analyzed (Participants) | 374
  HPV Type 11 | 79.9 [75.5 to 83.9]
  HPV Type 16: number analyzed (Participants) | 393
  HPV Type 16 | 94.9 [92.2 to 96.9]
  HPV Type 18: number analyzed (Participants) | 408
  HPV Type 18 | 40.2 [35.4 to 45.1]

20. Secondary Outcome: Geometric Mean Titers to HPV Types 6, 11, 16, and 18 at Month 120 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA)
Description: Antibodies to HPV types were measured using Luminex immunoassay (IgG-LIA). The unit of measure for this assay is IgG LIA mMU/mL; this unit cannot be directly compared with the cLIA mMU/mL unit reported for the cLIA results.
Time Frame: Month 120
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: IgG LIA mMU/mL
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
IgG LIA mMU/mL
  HPV Type 6: number analyzed (Participants) | 278
  HPV Type 6 | 38.8 [34.0 to 44.2]
  HPV Type 11: number analyzed (Participants) | 274
  HPV Type 11 | 31.0 [27.2 to 35.3]
  HPV Type 16: number analyzed (Participants) | 291
  HPV Type 16 | 162.0 [141.2 to 185.7]
  HPV Type 18: number analyzed (Participants) | 305
  HPV Type 18 | 19.7 [17.0 to 22.9]

21. Secondary Outcome: Percentage of Participants Seropositive for HPV Type 6, 11, 16, and 18 at Month 120 Assessed by IgG LIA
Description: Antibodies to HPV types were measured using IgG LIA. Thresholds for seropositive were ≥9, 6, 5, and 5 IgG LIA mMU/mL for HPV Types 6, 11, 16, and 18, respectively.
Time Frame: Month 120
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qHPV Vaccine in Base Study
Number analyzed (Participants) | 2025
Percentage of participants
  HPV Type 6: number analyzed (Participants) | 278
  HPV Type 6 | 91.7 [87.8 to 94.7]
  HPV Type 11: number analyzed (Participants) | 274
  HPV Type 11 | 92.0 [88.1 to 94.9]
  HPV Type 16: number analyzed (Participants) | 291
  HPV Type 16 | 99.7 [98.1 to 100]
  HPV Type 18: number analyzed (Participants) | 305
  HPV Type 18 | 92.1 [88.5 to 94.9]

ADVERSE EVENTS:
Time Frame: Base study: all AEs were collected systematically from Day 1 through Month 36. EXT 1: SAEs were collected systematically from Day 1 through Month 7. LTFU (EXT2): deaths and vaccine-related SAEs were collected up to 12 years after last dose of qHPV vaccine in Early Vaccination Group and up to 7 years after last dose of qHPV in Catch-up Vaccination Group.
Description: Medical Dictionary for Regulatory Activities (MedDRA) version 12.0 was used during the base study and follow-up, MedDRA version 14.1 was used during EXT1, and MedDRA version 20.0 was used during LTFU (EXT2).
  Participants at risk in EXT1 received ≥1 qHPV vaccination in EXT1 and had follow-up data.
  Other AEs were not solicited during EXT1 or LTFU (EXT2).
Groups:
- qHPV Vaccine: Base Study: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time participants received qHPV vaccination at Day 1, Month 2 and Month 6.
- Placebo: Base Study: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time participants received placebo at Day 1, Month 2 and Month 6.
- qHPV Vaccine: EXT1: Participants who received placebo and participants who received only 1 dose of qHPV vaccine in the base study were offered a complete 3-dose qHPV vaccine regimen (administered at EXT1 Day 1, Month 2 and Month 6). Participants who received only 2 doses of qHPV vaccine in the base study were offered a single additional dose of qHPV vaccine (administered at EXT1 Day 1).
- LTFU (EXT2): Participants received ≥1 dose of qHPV vaccine in Base Study, or received placebo in Base Study and qHPV vaccine in EXT1. This arm includes both groups enrolled in LTFU (EXT2): Early Vaccination Group and Catch-up Vaccination Group.
Arm/Group | qHPV Vaccine: Base Study | Placebo: Base Study | qHPV Vaccine: EXT1 | LTFU (EXT2)
All-Cause Mortality (participants affected / at risk) | 3/2020 | 10/2029 | 2/1084 | 7/1803
Serious Adverse Events (participants affected / at risk) | 8/2020 | 11/2029 | 3/1084 | 7/1803
Other Adverse Events (participants affected / at risk) | 1277/2020 | 1183/2029 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine: Base Study (N=2020) | Placebo: Base Study (N=2029) | qHPV Vaccine: EXT1 (N=1084) | LTFU (EXT2) (N=1803)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blast injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV Vaccine: Base Study (N=2020) | Placebo: Base Study (N=2029) | qHPV Vaccine: EXT1 (N=0) | LTFU (EXT2) (N=0)
Abdominal pain upper (Gastrointestinal disorders) | 19 (21) | 23 (23) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 40 (44) | 36 (38) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (30) | 16 (16) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 118 (131) | 125 (149) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 304 (446) | 275 (384) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 1116 (2087) | 992 (1767) | 0 (0) | 0 (0)
Injection Site Pruritus (General disorders) | 23 (27) | 24 (29) | 0 (0) | 0 (0)
Injection Site Swelling (General disorders) | 219 (318) | 187 (270) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 42 (43) | 44 (47) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 44 (46) | 50 (59) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 22 (23) | 20 (21) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 27 (28) | 20 (22) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 179 (222) | 207 (275) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 38 (38) | 37 (37) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.